CLINICAL TRIAL: NCT04620174
Title: Custom-made Versus Prefabricated Zirconia Crowns for Primary Molars; a Clinical Trial With 12-month Follow-up.
Brief Title: Custom-made Versus Prefabricated Zirconia Crowns for Primary Molars.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Roqaia Mohammad Alassar, Lecturer of Crowns and Bridges, Faculty of Dental Medicine for Girls, Al-Azhar University, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PD-P-020-006
Record Dates: First submitted 2020-11-03; First posted 2020-11-06 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Decayed Teeth
Keywords: Zirconia Crown, Primary teeth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Three groups will be included;
  1. Custom-made Zirconia Crowns Group (10 molars)
  2. Prefabricated Zirconia Crowns Group (10 molars)
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom-made zirconia crowns Group (Other): Ten decayed primary molars will be restored with custom-made zirconia crowns.
  Interventions: Other: Custom-made zirconia crowns
- Prefabricated zirconia crowns Group (Other): Ten decayed primary molars will be restored with prefabricated zirconia crowns.
  Interventions: Other: Prefabricated zirconia crowns

INTERVENTIONS:
Other: Custom-made zirconia crowns — Ten decayed primary molars will be restored with custom-made zirconia crowns.
  Arms: Custom-made zirconia crowns Group
Other: Prefabricated zirconia crowns — Ten decayed primary molars will be restored with prefabricated zirconia crowns.
  Arms: Prefabricated zirconia crowns Group

SUMMARY:
Background: Do construction methods of pediatric zirconia crowns affect the periodontal health and clinical performance of badly decayed primary molars? The question asked by many practitioners.

Purpose: to compare the periodontal health and clinical performance of primary molars restored with custom-made and prefabricated zirconia crowns. Hypothesis is the performance of primary molars restored with custom-made zirconia crowns will be equivalent to those restored with prefabricated zirconia crowns.

DETAILED DESCRIPTION:
This study is a randomized, 12-month follow up clinical trial. According to sample size calculation, ten patients will be selected in conjunction with departments of Pedodontics and Crowns & Bridges. The study will be conducted in accordance with the principles of the Research Ethics Committee, Faculty of Dental Medicine for Girls, Al-Azhar University, Egypt.

The purpose of the investigation and the clinical procedures of this study will be explained to the parents and children. A written informed consent form will be signed from patient guardians and obtained prior to study initiation. The inclusion and exclusion criteria are established as the following;

* Inclusion criteria

  1. Children of 5-9 years old.
  2. The children have at least 2 pulpotomized primary molars with no clinical signs & symptoms or periapical pathosis.
  3. Presence of an intact contralateral primary molar as a control.
  4. Willingness to participate and to continue with the follow up appointments.
  5. Clinical and radiographically confirmed dental caries extending to the middle third of dentin.
  6. Presence of teeth in opposite arch with normal occlusion.
* Exclusion criteria

  1. Children with systemic health problem.
  2. Children with periodontal disease.
  3. Children with unilateral chewing habit or allergic to local anesthesia.
  4. Presence of parafunctional habit.
* Clinical procedure;

  1. Patient selection and education; The participating children will continue with their routine dental appointments in the undergraduate training clinic. Before beginning, children, along with their parents will receive a standard oral hygiene education by an undergraduate student through brushing demonstration on a model. Parents will be warned when signs of gingival inflammation are present, or plaque control is inadequate.
  2. Samples grouping and teeth preparation:

     Forty primary molars will be included in the study. Twenty decayed teeth will be restored with crowns (10 with custom-made ZrCs and 10 with prefabricated ZrCs), and the other twenty intact contralateral teeth will be evaluated as the controls (10 molars will be the controls for custom-made ZrCs and 10 molars will be the controls for prefabricated ZrCs). Preparation of the crowns will be performed under local anesthesia, according to manufacturers' instructions with the following guidelines; 1-2mm occlusal reduction, 0.5-1mm axial reduction, and a chamfer finish line will be established 0.5-1mm subgingivally.
  3. Impression taking and temporization:

     After preparation, rubber-base impressions will be taken for the teeth specific for custom-made ZrCs. Then SSCs will be temporarily cemented over the prepared teeth till the next appointment.
  4. Try-in and cementation of ZrCs:

     SSCs will be removed and the custom-made and prefabricated ZrCs will be tried in and permanently cemented.
* Follow-up visits:

The participants will be recalled for evaluation after a baseline and at 1, 3, 6 and 12 months.

• Evaluation methods:

1. The periodontal health will be assessed using the plaque index (PI) and the gingival index (GI).
2. The clinical success of the crowns will be assessed in terms of crown retention, marginal adaptation, crown contour, fracture, stain resistance, opposing tooth wear and tooth exfoliation.

ELIGIBILITY:
Inclusion Criteria:

1. Children of 5-9 years old.
2. The children have at least 2 decayed primary molars.
3. Presence of an intact contralateral primary molar as a control.
4. Willingness to participate and to continue with the follow up appointments.
5. Clinical and radiographically confirmed dental caries extending to the middle third of dentin.
6. Presence of teeth in opposite arch with normal occlusion.

Exclusion Criteria:

1. Children with systemic health problem.
2. Children with periodontal disease.
3. Children with unilateral chewing habit or allergic to local anesthesia.
4. Presence of parafunctional habit.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change in periodontal health. | At 1, 3, 6 and 12 months following application.
  The periodontal health will be assessed using the plaque index (PI) and the gingival index (GI)

SECONDARY OUTCOMES:
Change in clinical performance. | At 1, 3, 6 and 12 months following application.
  The clinical success of the crowns will be assessed in terms of crown retention, marginal adaptation, crown contour, fracture, stain resistance, opposing tooth wear and tooth exfoliation.

CONTACTS AND LOCATIONS:
Overall Officials: Noha I Metwally, DDS, Principal Investigator — Pedodontist, Faculty of Dental Medicine for Girls, Al-Azhar University; Asmaa M Abdelgawad, DDS, Principal Investigator — Fixed Prosthodontist, Faculty of Dental Medicine for Girls, Al-Azhar University; Roqaia M Alassar, DDS, Principal Investigator — Fixed Prosthodontist, Faculty of Dental Medicine for Girls, Al-Azhar University
Locations (1):
- Roqaia M Alassar, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No